CLINICAL TRIAL: NCT03422497
Title: The Association of Sex With Provision of Guideline-based Perioperative Care for Hip Fracture Surgery Patients: a Population-based Study
Brief Title: The Association of Sex With Guideline-based Perioperative Care in Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM7
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Hip Fractures; Gender Bias; Surgery; Anesthesia
MeSH Terms: conditions — Hip Fractures; Sexism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male hip fracture surgery patients: Individuals 65 years or older admitted non-electively to hospital with a diagnosis of hip fracture who have surgery for their hip fracture and have male sex listed in their discharge abstract
  Interventions: Other: Male sex
- Female hip fracture surgery patients: Individuals 65 years or older admitted non-electively to hospital with a diagnosis of hip fracture who have surgery for their hip fracture and have female sex listed in their discharge abstract
  Interventions: Other: Female sex

INTERVENTIONS:
Other: Male sex — Male sex-as listed in the discharge abstract database
  Groups: Male hip fracture surgery patients
Other: Female sex — Male sex-as listed in the discharge abstract database
  Groups: Female hip fracture surgery patients

SUMMARY:
The investigators will use multilevel multivariable regression analysis to measure the association of sex with provision of guideline-based perioperative care for hip fracture surgery in Ontario.

DETAILED DESCRIPTION:
In 2013, the Ontario Ministry of Health and Longterm Care published a 'Quality Based Procedures' guideline for care of hip fracture patients. The adjusted association of sex with receipt of 5 perioperative processes of care that can be accurately measured in health administrative data within this guideline will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Non-elective hospital admission
* Hip fracture diagnosis
* Hip fracture surgery

Exclusion criteria

-None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Sex based on that listed in the discharge abstract database (not self-reported)
Study Population: Emergency hip fracture surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Perioperative geriatric medicine consult | Hospital admission to date of discharge from hospital, or 365 days after admission, whichever came first
  Physician billing code for perioperative, inpatient geriatric medicine consult or comprehensive assessment

SECONDARY OUTCOMES:
Preoperative anesthesiology consult | Hospital admission to date of surgery, or 365 days after admission, whichever came first
  Physician billing code for preoperative, inpatient anesthesiology consult
Wait for surgery greater than 2 days | Hospital admission to date of surgery, or 365 days after admission, whichever came first
  Hospital admission to surgery wait for greater than 2 days
Perioperative regional analgesia | Hospital admission to 3 days after surgery
  Peripheral nerve block or epidural administered in the perioperative period, identified from physician billing data codes
Neuraxial anesthesia | Day of surgery
  Spinal or epidural anesthesia, without concurrent general anesthesia, administered for the hip fracture surgery and identified from the discharge abstract database section which describes anesthesia techniques for surgery.

IPD SHARING:
Plan to Share IPD: No
Privacy policies in our institution preclude data sharing

REFERENCES:
- [Derived] Cho N, Boland L, McIsaac DI. The association of female sex with application of evidence-based practice recommendations for perioperative care in hip fracture surgery. CMAJ. 2019 Feb 11;191(6):E151-E158. doi: 10.1503/cmaj.180564. PMID 30745399